CLINICAL TRIAL: NCT03081364
Title: Patient Registry Of Magnetic Resonance Imaging in Non-Approved DEvices
Acronym: PROMeNADe
Status: Completed | Type: Observational
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 15-335
Record Dates: First submitted 2017-01-04; First posted 2017-03-16 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Magnetic Field Exposure
Keywords: Cardiac Implanted Device

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Outpatients: MRI; Critical Care Monitoring, Device Programming
  Interventions: Other: Initiate ACLS protocol if lethal arrythmia develops

INTERVENTIONS:
Other: Initiate ACLS protocol if lethal arrythmia develops — Cardiac Rhythm Management

SUMMARY:
The investigators are providing MRI in patients with non-MRI approved CIED's (Cardiac Implanted Electronic Devices)

DETAILED DESCRIPTION:
At Saint Luke's Hospital, despite growing evidence to the contrary, there is extremely limited data and experience with performing MRIs on patient with abandoned and epicardial leads in patients with non-approved ICDs and PMs. There is a limited mechanism to discuss this issue with the patient, screen the patient and assess their device beforehand, monitor them during the MRI examination, keep track of pulse sequences used, assess their devices after (and if necessary, resume prior programming before any changes), and to maintain that experience. The objective of this study is to create a protocol for an MRI at the commonly used magnetic strength of 1.5 T in patients that do not have conditional pacemakers and/or defibrillators and have abandoned or epicardial leads and maintain a registry of participants, devices involved, MRI examinations and pulse sequences used, and to keep records of any follow up events.

ELIGIBILITY:
Inclusion Criteria:

* Anyone with a cardiac device

Exclusion Criteria:

* Anyone who cannot consent for themselves or who don't have a durable power of attorney

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For all patients in whom a clinical MRI examination is felt to be important in the patients care, and in whom the potential benefits clearly outweigh the risks of an MRI exam as referred from various primary and/or subspecialty physicians.
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Change in Device Function | 3 years
  Change in lead impedance or sensing
Change in Thresholds of Pacing Lead | 3 years
  Measured in mA
Dysrhythmias Noted During Scan | 3 years
  Change in heart rhythm
Oxygen Saturation | 3 years
  Percentage of change or no change
Change in heart rate | 3 years
  Measured as beats per minute on single-lead heart monitor.
Patient Comments | 3 years
  Real-time patient report via intercom during scan of chest symptoms such as burning or aching
Interference Between the Implanted Cardiac Electronic Device and MRI | 3 years
  Measure any change in device battery voltage
Change in blood pressure | 3 years
  Monitored with automatic blood pressure cuff

CONTACTS AND LOCATIONS:
Overall Officials: Sanjaya K Gupta, MD, Principal Investigator — St. Luke's Hospital, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the IPD

REFERENCES:
- [Derived] Gupta SK, Ya'qoub L, Wimmer AP, Fisher S, Saeed IM. Safety and Clinical Impact of MRI in Patients with Non-MRI-conditional Cardiac Devices. Radiol Cardiothorac Imaging. 2020 Oct 22;2(5):e200086. doi: 10.1148/ryct.2020200086. eCollection 2020 Oct. PMID 33778621